CLINICAL TRIAL: NCT03420066
Title: NEXUS™ Aortic Arch Stent Graft System Data Collection Study for Compassionate-Use Procedures
Brief Title: The NEXUS™ Compassionate Use Data Collection Study
Status: Completed | Type: Observational
Sponsor: Endospan Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP008
Record Dates: First submitted 2018-01-28; First posted 2018-02-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Aortic Arch Aneurysm
MeSH Terms: conditions — Aneurysm, Aortic Arch

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective data collection: Group includes subjects that were implanted with the Nexus device as part of compassionate use procedure before joining the CIP008 study. Only intervention foreseen by CIP008 study is retrospective collection of data previously recorded as standard of care in medical charts (refer to Intervention/treatment section)
  Interventions: Other: Retrospective data collection

INTERVENTIONS:
Other: Retrospective data collection — Retrospective collection of data recorded as standard of care for patients that were implanted with the Nexus device as part of Compassionate Use duly authorized according to country specific regulations.

SUMMARY:
A Multicenter, observational Data Collection Study to Evaluate the Safety and Performance of the Nexus™ Aortic Arch Stent Graft System in patients that were implanted with the device as part of Compassionate Use Procedures.

DETAILED DESCRIPTION:
The purpose of the study is to collect and analyze data that is recorded as standard of care for patients that were implanted with the Nexus device as part of Compassionate Use Procedures.The data will be used to obtain additional information on the safety and performance of the Nexus™ Aortic Arch Stent Graft System in patients affected by pathologies involving the aortic arch.

Data will be collected at each time point of patient's follow up conducted according to the standard of care in each site.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom the Nexus implantation was initiated as part of a compassionate use procedure.
* A signed and dated Informed Consent document is available that authorizes to collect the patient's personal data following implantation of the Nexus systems and throughout the follow ups visits up to 5 years following implantation.

Exclusion Criteria:

-There are no exclusions. Data will be collected for all implanted population as described in the inclusion section above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will include all patients that were implanted with the Nexus device as part of the compassionate use.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Primary Safety Evaluation Criteria | within 30 days post implantation
  Device related mortality at 30 days post implantation based on review of medical charts by the Investigators
Performance Evaluation Criteria | within 30 days post implantation
  Successful disease treatment at 30 days post implantation, defined as Stent Graft positioned in the aortic arch isolating the diseased lesion based on review of medical charts by the Investigators.

SECONDARY OUTCOMES:
Secondary Safety Evaluation Criteria | within 1 year post-implantation
  Device related re-intervention (e.g. due to endoleak, stent graft occlusion, clinically significant migration) within 1 year from implantation and based on review of medical charts by the Investigators.

CONTACTS AND LOCATIONS:
Locations (4):
- Ospedale San Filippo Neri, Rome, Lazio, Italy
- ADHB Charitable Trust, Auckland, New Zealand
- Switzerland (2):
  - Klinik Hirslanden, Zurich
  - Zurich University Hospital, Zurich

IPD SHARING:
Plan to Share IPD: No